CLINICAL TRIAL: NCT00694720
Title: A Double-Blind, Randomized, Placebo-Controlled, Study Evaluating the Safety and Activity of Four Escalating Single Doses of AVE0657 in Congestive Heart Failure Patients Presenting as Cheyne-Stokes Breathing Syndrome
Brief Title: Evaluation of the Effect of AVE0657 in Cheynes-Stokes Breathing Syndrome Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination following reassessment of the potential benefit-risk of AVE0657
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT6795; EudraCT 2007-002172-34
Record Dates: First submitted 2008-05-07; First posted 2008-06-10 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Heart Failure; Sleep Apnea Syndromes; Cheyne-Stokes Respiration
Keywords: Cheyne-stokes breathing
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes; Cheyne-Stokes Respiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dose Level 1 (Experimental)
  Interventions: Drug: AVE0657
- Dose Level 2 (Experimental)
  Interventions: Drug: AVE0657
- Dose Level 3 (Experimental)
  Interventions: Drug: AVE0657
- Dose Level 4 (Experimental)
  Interventions: Drug: AVE0657
- Placebo (Placebo Comparator): 12 subjects: 3 subjects per dose level
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AVE0657 — capsules once a day at bedtime
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4
Drug: placebo — capsules once a day at bedtime
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the activity on breathing parameters of 4 escalating doses of AVE0657 in comparison to placebo in patients with Cheynes-Stokes Breathing Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Congestive heart failure (CHF) defined as ejection fraction ≤40% by history of echocardiography data and New York heart Association (NYHA) class II-III and of typical cyclic crescendo and decrescendo change in breathing amplitude AHI ≥10 and <60 and majority of the apneas to be ≥60% central in origin.

Exclusion Criteria:

* Subject on supplemental oxygen

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change in the Apnea Hypopnea Index (AHI) | 2 days

SECONDARY OUTCOMES:
Safety and tolerability | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick LEVY, Professor, Principal Investigator — Hôpital Michallon - Grenoble - France
Locations (3):
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Barcelona, Spain